CLINICAL TRIAL: NCT05109533
Title: Probiotics Role in HPV Clearance When Coexisting Vaginal Infections
Brief Title: Probiotics Role in HPV Cervico-vaginal Infection Clearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Lavinia Domenici, Principal Investigator, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3644
Record Dates: First submitted 2021-08-17; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Vaginal Infection; HPV Infection
Keywords: vaginal infections; probiotics; HPV
MeSH Terms: conditions — Vaginitis; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - ARM WITH STANDARD TREATMENT (No Intervention): Standard specific treatment for vaginal infections following latest version of CDC guidelines
- Group 2 - ARM WITH STANDARD TREATMENT PLUS PROBIOTICS IMPLEMENTATION (Experimental): Standard specific treatment for vaginal infections plus long-lasting (9 months) vaginal and oral probiotics implementation (Lactobacillus rhamnosus BMX 54 vaginally and Lactobacillus reuteri RC-14/Lactobaciullus rhamnosus GR-1 combination orally)
  Interventions: Other: Lactobacillus rhamnosus BMX 54, Lactobacillus reuteri RC-14, Lactobacillus rhamnosus GR-1

INTERVENTIONS:
Other: Lactobacillus rhamnosus BMX 54, Lactobacillus reuteri RC-14, Lactobacillus rhamnosus GR-1 — Probiotics implementation
  Arms: Group 2 - ARM WITH STANDARD TREATMENT PLUS PROBIOTICS IMPLEMENTATION

SUMMARY:
Vaginal infections demonstrated to be implicated in the persistence of HPV, activating a vicious circle of vaginal microbial perturbations. HPV infection can destroy the biofilm barrier formed by the local vaginal immune microenvironment, leading to a condition called dysbiosis. Contemporarily, the resulting local microecological imbalance in the vagina can subsequently upregulate the expression of the HPV protein, increasing HPV-related cytological alterations.

DETAILED DESCRIPTION:
A total of 483 women affected by different vaginal infections and concomitant HPV-positivity were enrolled between 2018 and 2020 at Department of Gynecological, Obstetrical and Urological Sciences, University "Sapienza" of Rome (Rome, Italy) and 2nd Division of Obstetrics and Gynecology, Azienda Ospedaliera Universitaria Pisana, University of Pisa (Pisa, Italy). Women with positive swabs for infections were randomized in two groups, standard specific treatment (n=231) versus the standard treatment plus long-lasting (9 months) vaginal and oral probiotics implementation (n=252).

ELIGIBILITY:
Inclusion criteria

* age > 18 years
* positive swabs for vaginal infections detected during colposcopy check
* HPV test positivity

Exclusion Criteria:

* pregnancy or breastfeeding
* concomitant malignancies
* immunological diseases
* severe comorbidities
* prolonged corticosteroid treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Vaginal infection as inclusion criteria
Enrollment: 483 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of a possible role of probiotics in HPV clearance | 12 months
  Changes in HPV test positivity
Evaluation in vaginal infection resolution | 12 months
  Negative swab test for vaginal infections, complete symptoms resolution, absence of colposcopy findings suggestive for permanence of infections (e.g. colpitis, fine punctuation, etc), absence of infection following Amsel's criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Domenici L. Letter to "The application of PAX1 methylation detection and HPV E6/E7 mRNA detection in cervical cancer screening". J Obstet Gynaecol Res. 2021 Sep;47(9):3419-3420. doi: 10.1111/jog.14912. Epub 2021 Jun 21. No abstract available. PMID 34155727
- [Background] Palma E, Recine N, Domenici L, Giorgini M, Pierangeli A, Panici PB. Long-term Lactobacillus rhamnosus BMX 54 application to restore a balanced vaginal ecosystem: a promising solution against HPV-infection. BMC Infect Dis. 2018 Jan 5;18(1):13. doi: 10.1186/s12879-017-2938-z. PMID 29304768
- [Background] Recine N, Palma E, Domenici L, Giorgini M, Imperiale L, Sassu C, Musella A, Marchetti C, Muzii L, Benedetti Panici P. Restoring vaginal microbiota: biological control of bacterial vaginosis. A prospective case-control study using Lactobacillus rhamnosus BMX 54 as adjuvant treatment against bacterial vaginosis. Arch Gynecol Obstet. 2016 Jan;293(1):101-107. doi: 10.1007/s00404-015-3810-2. Epub 2015 Jul 5. PMID 26142892